CLINICAL TRIAL: NCT04268615
Title: Covert Saccade Triggers in Bilateral Vestibular Hypofunction
Acronym: CS-TRIGGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0998; 2020-A00184-35 (Other: ID-RCB)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2022-07

CONDITIONS: Reflex, Abnormal; Bilateral Vestibulopathy; Healthy Volunteers
Keywords: Saccadic Eye Movements; Bilateral Vestibulopathy; Bilateral Vestibular Hypofunction
MeSH Terms: conditions — Reflex, Abnormal; Bilateral Vestibulopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Experimental): Patients suffering from chronic bilateral vestibular hypofunction
  Interventions: Other: Covert Saccades and Virtual Reality; Other: Actives versus passives Head Impulses; Other: Visually guided saccades
- healthy subject group (Active Comparator)
  Interventions: Other: Covert Saccades and Virtual Reality; Other: Actives versus passives Head Impulses; Other: Visually guided saccades

INTERVENTIONS:
Other: Covert Saccades and Virtual Reality — During this intervention, patients will undergo head impulse testing while wearing virtual reality Headsets. During the head impulse tests the visual information will be modified in order to create a conflict between head rotation and rotation of the visual scene. Recording of head and eye movement will be done during these head impulses in order to verify if visual information modifies compensatory eye movements during head impulses.
Other: Actives versus passives Head Impulses — Patients will undergo classic passive head rotation as well as active head rotation in order to compare latencies of covert saccades in both conditions.
Other: Visually guided saccades — Patients as well as healthy control subjects will undergo testing of visually guided saccades in different conditions (step, gap, overlap) in order to compare latencies of covert saccades between both groups.

SUMMARY:
Patients with chronic bilateral vestibular hypofunction may suffer from a visual instability during head movement called oscillopsia. Visual consequence of vestibular deficit can lead to a severe impairment of their quality of life. However, correcting saccades during rapid head movement, called covert-saccades, have been more recently identified. These saccades, which occur during the head movement in patients with vestibular hypofunction, present a very short latency. They could compensate for the lack of vestibular-ocular reflex and greatly decrease oscillopsia and visual impairment. The triggering of these covert-saccade is still not known. They could be of visual origin but the short latency is unusual. The objective of this study is to evaluate the potential role of visual trigger in 12 patients with chronic bilateral areflexia, using different visuo-vestibular conditions. The latency of simple visually guided saccades will also be tested in the group of patients and a group of 12 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* For all :

  * Age from 18 to 90
  * Understanding of the experimental instructions
  * Informed Consent
* For Patients :

Bilateral vestibular hypofunction with regards to the criteria of the of the Barany Society A. Chronic vestibular syndrome with at least three of the following symptoms

1. Postural imbalance
2. Unsteadiness of gait
3. Movement-induced blurred vision or oscillopsia during walking or quick head/body movements
4. Worsening of postural imbalance or unsteadiness of gait in darkness and/or on uneven ground B. No symptoms while sitting or lying down under static conditions C. Bilaterally reduced or absent angular VOR function documented by

   * bilaterally pathological horizontal angular VOR gain < 0.6, measured by the video-HIT5or scleral-coil technique and/or
   * reduced caloric response (sum of bithermal max. peak SPV on each side < 6°/sec7)and/or
   * reduced horizontal angular VOR gain < 0.1 upon sinusoidal stimulation on a rotatorychair (0.1 Hz, Vmax = 50°/sec).

D. Not better accounted for by another disease

* For Healthy control No ENT or neurological disorders

Exclusion Criteria:

* Corrected Visual Acuity lower than 5/10
* Other conditions leading to oscillopsia or ataxia
* Oculomotor palsy, ocular instability in primary position
* Treatment that may affect ocular motility (psychotropes)
* Cervical rachis pathology with instability
* Cochlear Implants
* Non-stabilized medical disease
* Pregnant women
* Patients under tutelage
* Patient without social security

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Latency of covert-saccades | Day 1
  Latency of covert saccades correspond to the time between the beginning of head impulse and the initiation of the first covert-saccade

SECONDARY OUTCOMES:
Frequency of covert-saccades | Day 1
  Frequency of covert saccades corresponds to the total amount of covert-saccades divided by the total amount of head impulse tests multiplied by 100.
Velocity of covert-saccades | day 1
  Velocity of covert saccades correspond to the maximal velocity of the first covert-saccade
Amplitude of covert-saccades | Day 1
  Amplitude of covert saccades correspond to amplitude of the first covert-saccade
Latency of visually-guided saccades | Day 1
  Latency of visually guided saccades correspond to the time between the appearance of target and the initiation of the first saccade

CONTACTS AND LOCATIONS:
Overall Officials: Caroline FROMENT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lagadec V, Pelisson D, Koun E, Robert C, Froment Tilikete C, Hermann R. Oculomotor compensatory strategies in bilateral vestibulopathy: Predictive and active conditions of head movements. J Vestib Res. 2025 Nov;35(6):290-299. doi: 10.1177/09574271251355180. Epub 2025 Jun 21. PMID 40543046
- [Background] Hermann R, Ramat S, Colnaghi S, Lagadec V, Desoche C, Pelisson D, Froment Tilikete C. Catch-Up Saccades in Vestibulo-Ocular Reflex Deficit: Contribution of Visual Information? Ear Hear. 2025 May-Jun 01;46(3):719-728. doi: 10.1097/AUD.0000000000001616. Epub 2024 Dec 18. PMID 39690450
- [Background] Desoche C, Verdelet G, Salemme R, Farne A, Pelisson D, Froment C, Hermann R. Virtual reality set-up for studying vestibular function during head impulse test. Front Neurol. 2023 Mar 29;14:1151515. doi: 10.3389/fneur.2023.1151515. eCollection 2023. PMID 37064179